CLINICAL TRIAL: NCT07236541
Title: Impact of Airway Mucus Plugs on Secondary Pulmonary Fibrosis in COPD Patients: A Single-Center Case-Control Study
Status: Recruiting | Type: Observational
Sponsor: Ming Zhong (Other)
Responsible Party: Sponsor-Investigator, Ming Zhong, Chief Physician and Professor, Department of Pulmonary and Critical Care Medicine, Zhongshan Hospital, Fudan University, Shanghai Zhongshan Hospital
Organization: Shanghai Zhongshan Hospital (Other)
Other Study IDs: B2025-657
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Lung Fibrosis
MeSH Terms: conditions — Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COPD（chronic hypoxia）
  Interventions: Other: No intervention; observational biospecimen collection only
- Normal（Normoxia）
  Interventions: Other: No intervention; observational biospecimen collection only

INTERVENTIONS:
Other: No intervention; observational biospecimen collection only — No intervention; observational biospecimen collection only

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is frequently accompanied by airway mucus plugs, which are closely associated with airflow obstruction, acute exacerbations, and increased mortality. However, whether mucus plugs contribute to secondary pulmonary fibrosis remains unclear. This single-center, prospective, case-control study aims to investigate the relationship between airway mucus plugs and lung fibrosis in patients with COPD undergoing lung cancer surgery.

During surgery, distal non-tumorous lung tissues and airway mucus will be collected for histological and molecular analyses. Mucus plug burden will be quantified using AB-PAS staining, and fibrosis will be assessed using Masson staining. Expression of epithelial-mesenchymal transition (EMT) markers, fibrotic markers, and the mechanosensitive ion channel Piezo1 will also be measured. COPD patients (FEV₁/FVC <0.70) will be compared with non-COPD surgical controls.

The study aims to clarify whether mucus plugs are associated with increased fibrosis and to explore the potential involvement of mechanical-signaling pathways, including Piezo1 activation. Findings may provide new clinical and pathological evidence for mucus-induced fibrotic remodeling in COPD and help identify novel therapeutic targets.

ELIGIBILITY:
Inclusion Criteria:

* ① Age ≥ 18 years old;

  * Planned radical resection for lung cancer, with postoperative pathological diagnosis of primary lung cancer;

    * During surgery, non tumor lung tissue at a distance of ≥ 5 cm from the tumor edge can be obtained; ④ Case group: Preoperative pulmonary function examination confirmed diagnosis of COPD (FEV ₁/FVC<0.70); ⑤ Control group: Preoperative lung function was normal (FEV ₁/FVC ≥ 0.70), with no history of COPD; ⑥ The subjects are able to understand and sign the informed consent form

Exclusion Criteria:

* ① Clear presence of other interstitial lung diseases (ILD) or idiopathic pulmonary fibrosis before or during surgery （IPF）、 Fibrosis after pneumoconiosis or tuberculosis;

  * Active pulmonary infections (such as bacterial pneumonia, fungal infections, active tuberculosis);

    * Having received neoadjuvant radiotherapy or chemotherapy, which may affect the morphology or molecular results of distal lung tissue; ④ Combined severe immunodeficiency or long-term systemic immunosuppressive therapy (such as glucocorticoids ≥ 20 mg/d, More than 4 weeks);

      * Merge with other serious systemic diseases (such as advanced heart failure, end-stage renal disease), affecting study compliance or Survival expectation; ⑥ Pregnant or lactating women; ⑦ Refusing to sign the informed consent form or deemed unsuitable by the researcher to participate in the study.

Ages: 18 Years to 89 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients undergoing lung cancer surgery at Zhongshan Hospital, Fudan University. Participants include two groups: (1) patients with chronic obstructive pulmonary disease (COPD), defined by a pre-operative post-bronchodilator FEV₁/FVC <0.70; and (2) non-COPD surgical controls with normal lung function. During clinically indicated lung cancer resection, distal non-tumorous lung tissue samples and airway mucus (if present) are collected without adding any additional surgical risk. All participants are ≥18 years old and able to provide informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-10-30 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Clarify the relationship between airway mucus embolism and secondary pulmonary fibrosis in COPD patients | At the time of surgery and within 6 months after sample collection for laboratory analysis
  By comparing the distal lung tissue of patients undergoing COPD and non COPD lung cancer surgery, a systematic evaluation was conducted to determine the difference between airway mucus thrombus load and the degree of lung tissue fibrosis, and to answer whether airway mucus thrombus is an important pathological factor promoting secondary pulmonary fibrosis in COPD.

SECONDARY OUTCOMES:
The correlation between mucus plugs and clinical features | At the time of surgery and within 6 months after sample collection for laboratory analysis
  Explore the relationship between mucus clot burden and clinical characteristics (such as smoking history, lung function, hypoxic status) and pathological indicators of patients.
  The association between mucus plugs and fibrosis molecular markers:
  Detect and compare epithelial mesenchymal transition (EMT) related molecules (E-cadherin, Vimentin), fibrosis markers (α - SMA, COL1A1), inflammatory markers, etc., to clarify the association between mucosal thrombus load and molecular level fibrosis response.
  Possible functions of Piezo1 channel:
  Preliminary exploration of the correlation between mucus clot load and Piezo1 expression and activity, providing clinical pathological evidence for revealing the role of mechanical pathways in mucus induced fibrosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No